CLINICAL TRIAL: NCT03587142
Title: Buspirone for Early Satiety and Symptoms of Gastroparesis: A Multicenter, Randomized, Placebo-Controlled, Double-Masked Trial (BESST)
Brief Title: Buspirone for Early Satiety and Symptoms of Gastroparesis
Acronym: BESST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Texas Tech University Health Sciences Center, El Paso (Other); Johns Hopkins University (Other); Temple University (Other); University of Louisville (Other); Wake Forest University (Other); Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10- GpCRC3-BESST; U01DK073983 (NIH); U01DK112193 (NIH); U01DK073975 (NIH); U01DK074035 (NIH); U01DK074007 (NIH); U01DK073974 (NIH); U24DK074008 (NIH)
Record Dates: First submitted 2018-07-02; First posted 2018-07-16 (Actual); Results first posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Gastroparesis
Keywords: gastroparesis; early satiety; stomach; buspirone; 5-HT 1a receptor agonist
MeSH Terms: conditions — Gastroparesis | interventions — Buspirone

STUDY DESIGN:
Intervention Model Description: BESST is a multi-center, randomized, placebo-controlled, double-masked, parallel treatment groups phase 2 trial with half the participants receiving the study drug, buspirone, and half receiving the placebo.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants, all clinic staff and the investigators will be masked as to whether the participant is receiving buspirone or the placebo.
  The study drug will be over encapsulated in a size 0 gelatin capsule with partial filler to be identical to the placebo capsule, which contains only filler.
  The random treatment assignment will consist of a numbered study drug bottle; each bottle number will be unique and each participant will be assigned a specific bottle number, which is labelled: "Buspirone or placebo 10 mg." with directions.
  The randomization scheme will assign participants in randomly permuted blocks of assignments stratified by clinical center. The randomization plan will be prepared and administered centrally via a secure web application by the Scientific Data Research Center.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Buspirone (Active Comparator): Buspirone HCl 10 mg capsule orally three times daily, 30 minutes before each meal, for 4-weeks
  Interventions: Drug: Buspirone
- Placebo (Placebo Comparator): Placebo capsule orally three times daily, 30 minutes before each meal, for 4-weeks; manufactured to look identical to buspirone capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Buspirone — Buspirone tablet
  Other Names: Buspar; buspirone hydrochloride (HCl); Buspar Dividose; Vanspar
  Arms: Buspirone
Drug: Placebo — "Sugar" pill manufactured to mimic buspirone 10 mg tablet
  Other Names: Placebo (for buspirone)
  Arms: Placebo

SUMMARY:
This study evaluates whether the study medication, buspirone, an antianxiety drug, improves the symptoms of gastroparesis in patients with gastroparesis symptoms and at least moderately severe symptoms of fullness and/or inability to eat a full meal. Half the patients will receive buspirone and half the patients will receive a placebo.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-masked, placebo-controlled, parallel treatment groups phase 2 trial to determine the effect of buspirone, a 5-hydroxytryptamine (5-HT) 1a receptor agonist, on early satiety and postprandial fullness in participants with symptoms of gastroparesis and with at least moderately severe symptoms of early satiety and/or postprandial fullness. After enrollment, participants aged 18-75 years will be treated with buspirone (10 mg three times per day) or a matching placebo for 4 weeks, followed by a 2-week post-treatment washout period. The primary outcome for the study is 4-week change (week 4 minus baseline) in the 4-item postprandial fullness/early satiety subscore (higher scores indicate worse symptoms) from the Patient Assessment of Gastrointestinal Disorders Symptom Severity Index (PAGI-SYM) Gastroparesis Cardinal Symptom Index (GCSI). We hypothesize that buspirone treatment will improve symptoms of postprandial fullness/early satiety compared to treatment with placebo, as indicated by a lower (smaller, more negative) 4-week change in the postprandial fullness/early satiety subscore in the buspirone arm compared to the placebo arm; change for a participant will be calculated as subscore at 4-weeks minus subscore at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 85 years of age at initial screening interview
* Symptoms compatible with gastroparesis or other functional gastric disorder for at least 3 months (does not have to be contiguous) prior to initial screening interview
* Diagnosis of either diabetic or idiopathic gastroparesis
* Delayed or normal gastric emptying retention on screening 4-hour Gastric Emptying Scintigraphy test
* Symptoms of gastroparesis measured by the 9-item PAGI-SYM Gastroparesis Cardinal Symptom Index (GCSI) total score > 2.0 at enrollment
* Symptomatic with postprandial fullness/early satiety severity at enrollment using the PAGI-SYM GCSI post-prandial fullness/early satiety subscore ≥ 3
* Upper endoscopy or upper GI series without ulcers or mass lesions in the 2 years prior to enrollment

Exclusion Criteria:

* Post-surgical gastroparesis, including prior pyloromyotomy, pyloric resection, vagotomy, bariatric surgery or post-Nissen fundoplication
* Another active disorder which could explain symptoms in the opinion of the investigator
* Concurrent use of opiate narcotic analgesics more than 3 days per week
* Significant hepatic injury as defined by alanine aminotransferase (ALT) elevation of greater than twice the Upper Limit of Normal (ULN) or a Child-Pugh score of 10 or greater
* Significant renal impairment as defined by serum creatinine > 3.0
* Uncontrolled diabetes defined as HbA1c (%) of 10% or more within 60 days of enrollment
* Allergy to buspirone
* Concurrent or prior use (within 30 days) of monoamine oxidase (MAO) inhibitors
* Concurrent or prior use (within 30 days) of benzodiazepines
* Concurrent or prior use (within 30 days) of buspirone, warfarin, haloperidol, and drugs to treat seizures (e.g., phenytoin and carbamazepine)
* Women breast feeding or known to be pregnant
* Any other condition, which in the opinion of the investigator would impede compliance or hinder completion of the study
* Failure to give informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2019-08-27 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry P Parkman, MD, Principal Investigator — Temple University Hospital, Philadelphia, PA; Pankaj J Pasricha, MD, Study Chair — Johns Hopkins Hospital, Baltimore, MD
Locations (6):
- United States (6):
  - University of Louisville, Louisville, Kentucky
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Temple University, Philadelphia, Pennsylvania
  - Texas Tech University Health Science Center, El Paso, Texas

IPD SHARING:
Plan to Share IPD: Yes
The study will comply with the NIH Data Sharing Policy. The data will be first de-identified so that no individual participant identifiers will be included in the dataset (no names, addresses, dates, comments, etc). If a characteristic is an extreme value for this population, then those values will be categorized into one frequency group. If a CSR has multiple versions, then all data will be recoded into the format of the most current form version. A random unique identification number will be substituted for the unique BESST identification number. If a clinical item was obtained from surveys with restrictions due to licensing, then that data will be excluded. The data will be shared in 2 stages: the first will be the analytic datasets to produce the primary outcome paper. For this dataset, the documentation will include analytic code. The full dataset by CSR will be provided in the second stage.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The analytic datasets to produce the primary result manuscript will be submitted within one year of publication of the primary result manuscript. The full clinical dataset for all Clinical Study Reports (CSRs) without proprietary restrictions will be submitted within 2 years of the primary result manuscript publication. This data will be available publicly indefinitely.
Access Criteria: An investigator interested in acquiring BESST study data should contact the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) Central Repository at https://www.niddkrepository.org/search/study/ and apply to obtain the data required for their study.
URL: https://repository.niddk.nih.gov/home/

REFERENCES:
- See also: Link to the Gastroparesis Clinical Research Consortium (GpCRC) web site Home page. There are some open-links for patients, such as Information for Patients. — https://jhuccs1.us/gpcrc/default.asp

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 131 adult participants with gastroparesis or gastroparesis-like 28, symptoms with at least moderately severe symptoms of early satiety and post-prandial fullness and a normal endoscopy were recruited at 6 tertiary clinic sites located in the U.S. between August 2019 and February 2022. The first participant was enrolled August 27, 2019 and the last participant was enrolled February 28, 2022.
Pre-assignment Details: Of the 131 participants assessed for eligibility, 96 met eligibility criteria and provided informed consent and were randomized to treatment (47 to Buspirone arm and 49 to Placebo arm).
Period: Overall Study
Arm/Group | Buspirone | Placebo
Started | 47 | 49
Completed | 39 | 39
Not Completed | 8 | 10
Not completed — Lost to Follow-up | 5 | 3
Not completed — Did not complete the f4 visit | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Buspirone | Placebo | Total
Number analyzed (Participants) | 47 | 49 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.0 (15.8) | 44.2 (15.0) | 43.6 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 45 | 88
  Male | 4 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 17 | 30
  Not Hispanic or Latino | 34 | 32 | 66
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 5 | 7
  White | 43 | 41 | 84
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1
Married [Count of Participants; unit: Participants] — Marital status: married or not married
  Participants | 16 | 21 | 37
Diabetes Type 1 [Count of Participants; unit: Participants] — Diagnosed with Diabetes, Type 1 at baseline: Yes or no.
  Participants | 3 | 6 | 9
Diabetes Type 2 [Count of Participants; unit: Participants] — Diagnosed with Diabetes Type 2 at baseline: Yes vs no.
  Participants | 13 | 15 | 28
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.5 (7.5) | 29.8 (7.3) | 29.7 (7.4)
Overweight to obese (BMI>/=25 kg/m^2) [Count of Participants; unit: Participants] | 31 | 37 | 68
Weight [Mean (Standard Deviation); unit: kilogram] | 78.1 (21.2) | 80.2 (22.2) | 79.2 (21.6)
Waist circumfence [Mean (Standard Deviation); unit: centimeter] | 98.1 (22.2) | 98.2 (19.6) | 98.1 (20.8)
Proton pump inhibitors [Count of Participants; unit: Participants] | 35 | 34 | 69
Anxiolytic [Count of Participants; unit: Participants] | 1 | 0 | 1
Antiemetic [Count of Participants; unit: Participants] | 31 | 25 | 56
Narcotic (3X/week or less) [Count of Participants; unit: Participants] | 2 | 4 | 6
Anti-depressant [Count of Participants; unit: Participants] | 22 | 22 | 44
Neuropathic or pain modulator, anti-seizure, or other psychiatric medication [Count of Participants; unit: Participants] | 28 | 31 | 59
Gastroparesis Cardinal Symptom Index (GCSI), total score [Mean (Standard Deviation); unit: units on a scale] — The 9-item Gastroparesis Cardinal Symptom Index (GCSI) total score rates gastroparesis symptom severity in the prior 2 weeks, determined by averaging 3 subscores: Nausea/Vomiting (average of 3 items: nausea, vomiting, retching), the Early Satiety/ Postprandial Fullness subscore (average of 4 items (stomach fullness, inability to finish a meal, feeling excessively full after meals, and loss of appetite) and the bloating subscore which is average of 2 items (bloating, stomach distention). The scale ranges from 0 to 5, where 0 is no symptoms and 5= very severe symptoms.
  units on a scale | 3.6 (0.7) | 3.5 (0.6) | 3.5 (0.6)
Nausea/vomiting subscale [Mean (Standard Deviation); unit: units on a scale] — This subscale from the Gastroparesis Cardinal Index (GCSI) survey is the average of severity in the prior 2 weeks of nausea, vomiting, and retching symptoms on a scale of 0 to 5, where 0=none and 5=very severe symptoms.
  units on a scale | 2.5 (1.3) | 2.4 (1.3) | 2.5 (1.3)
Nausea severity [Mean (Standard Deviation); unit: units on a scale] — This is 1 item of the Gastroparesis Cardinal Index (GCSI) survey rating the severity of nausea on a scale from 0 (none) to 5 (very severe).
  units on a scale | 3.6 (1.3) | 3.6 (1.2) | 3.6 (1.3)
Retching severity [Mean (Standard Deviation); unit: units on a scale] — This is 1 item of the Gastroparesis Cardinal Index (GCSI) survey rating the severity of retching in the prior 2-weeks on a scale from 0 (none) to 5 (very severe).
  units on a scale | 2.1 (1.7) | 1.8 (1.6) | 2.0 (1.6)
Vomiting severity [Mean (Standard Deviation); unit: units on a scale] — This is 1 item of the Gastroparesis Cardinal Index (GCSI) survey rating the severity of vomiting in the prior 2-weeks on a scale from 0 (none) to 5 (very severe).
  units on a scale | 1.9 (1.8) | 1.8 (1.7) | 1.8 (1.7)
Fullness/early satiety subscale [Mean (Standard Deviation); unit: units on a scale] — This measure is the average of early satiety/postprandial fullness symptom severity in the prior 2-weeks, comprised of 4 items on the Gastroparesis Cardinal Symptom (GCSI) inventory: the average of stomach fullness, inability to finish a normal-sized meal, feeling excessively full after meals, and loss of appetite symptom scores; rated on a scale of 0 (no symptoms) to 5 (very severe symptoms).
  units on a scale | 4.0 (0.6) | 4.0 (0.6) | 4.0 (0.6)
Stomach fullness severity [Mean (Standard Deviation); unit: units on a scale] — This is 1 item of the Gastroparesis Cardinal Index (GCSI) survey rating the severity of stomach fullness in the prior 2 weeks on a scale from 0 (none) to 5 (very severe).
  units on a scale | 4.2 (0.8) | 4.2 (0.7) | 4.2 (0.7)
Unable to finish meal severity [Mean (Standard Deviation); unit: units on a scale] — This is 1 item of the Gastroparesis Cardinal Index (GCSI) survey rating the severity of the inability to finish a normal sized meal in the prior 2 weeks on a scale from 0 (none) to 5 (very severe).
  units on a scale | 4.0 (1.0) | 4.0 (0.9) | 4.0 (0.9)
Excessive fullness severity [Mean (Standard Deviation); unit: units on a scale] — This is 1 item of the Gastroparesis Cardinal Index (GCSI) survey rating the severity of excessive fullness in the prior 2 weeks on a scale from 0 (none) to 5 (very severe).
  units on a scale | 4.2 (0.9) | 4.3 (0.7) | 4.3 (0.8)
Loss of appetite severity [Mean (Standard Deviation); unit: units on a scale] — This is 1 item of the Gastroparesis Cardinal Index (GCSI) survey rating the severity of loss of appetite in the prior 2 weeks on a scale from 0 (none) to 5 (very severe).
  units on a scale | 3.6 (1.3) | 3.5 (1.2) | 3.5 (1.2)
Bloating subscale [Mean (Standard Deviation); unit: units on a scale] — This is comprised of the average of 2 items (bloating, stomach or belly visibly larger on the Gastroparesis Cardinal Index (GCSI) survey rating the severity of average bloating symptoms the prior 2 weeks on a scale from 0 (none) to 5 (very severe).
  units on a scale | 4.2 (1.0) | 3.9 (1.0) | 4.1 (1.0)
Bloating severity [Mean (Standard Deviation); unit: units on a scale] — This is 1 item of the Gastroparesis Cardinal Index (GCSI) survey rating the severity of bloating in the prior 2 weeks on a scale from 0 (none) to 5 (very severe).
  units on a scale | 4.4 (0.9) | 4.0 (1.1) | 4.2 (1.0)
Stomach distention severity [Mean (Standard Deviation); unit: units on a scale] — This is 1 item of the Gastroparesis Cardinal Index (GCSI) survey rating the severity of stomach distention or visibly larger belly or stomach in the prior 2 weeks on a scale from 0 (none) to 5 (very severe).
  units on a scale | 4.0 (1.2) | 3.9 (1.1) | 4.0 (1.1)
Upper abdominal pain subscale [Mean (Standard Deviation); unit: units on a scale] — This is the average of 2 items, upper abdominal (above the navel) pain, Upper abdominal (above the navel) discomfort, on the Patient assessment of upper gastrointestinal symptom severity index (PAGI-SYM) survey rating the severity of upper abdominal pain/discomfort in the prior 2 weeks on a scale from 0 (none) to 5 (very severe).
  units on a scale | 3.3 (1.3) | 3.0 (1.2) | 3.1 (1.2)
Gastroesophageal Reflux (GERD) subscale [Mean (Standard Deviation); unit: units on a scale] — This is the average of 7 items: Heartburn during the day; heartburn while lying down; regurgitation (fluid or liquid from your stomach coming up into your throat) during the day; regurgitation while lying down; feeling of discomfort inside your chest during the day; feeling of discomfort during sleep time; bitter, acid or sour taste in your mouth, on the Patient assessment of upper gastrointestinal symptom severity index (PAGI-SYM) survey rating the severity of gastroesophageal reflux symptoms (GERD) in the prior 2 weeks on a scale from 0 (none) to 5 (very severe).
  units on a scale | 2.1 (1.4) | 2.3 (1.2) | 2.2 (1.3)
Predominant symptom cluster [Count of Participants; unit: Participants]
  Excessive fullness | 4 | 13 | 17
  Early satiety or loss of appetite | 2 | 4 | 6
  Bloating or distended stomach | 14 | 10 | 24
  Nausea or vomiting or retching | 15 | 13 | 28
  Upper abdominal pain or discomfort | 5 | 1 | 6
  Lower abdominal pain or discomfort | 4 | 1 | 5
Gastrointestinal Symptom Rating Scale (GSRS) [Mean (Standard Deviation); unit: units on a scale] — The 15-item disease-specific Gastrointestinal Symptom Rating Scale (GSRS) total score is an average 5 symptom clusters: Reflux, Abdominal pain, Indigestion, Diarrhoea and Constipation; each item is rated not (0) to very severe discomfort (7) of the symptom in the past week.
  units on a scale | 3.8 (1.0) | 3.7 (1.1) | 3.8 (1.0)
Patient Health Questionnaire somatization severity scale (PHQ-15) [Mean (Standard Deviation); unit: units on a scale] — The Patient Health Questionnaire somatization severity scale (PHQ-15) total score is comprised of 15 somatic symptoms rated from 0 (not) to 2 (very bothered a lot) in the prior 4 weeks, ranging from 0 to 30 where 30 is very severe level of somatization.
  units on a scale | 14.7 (5.0) | 14.9 (4.1) | 14.8 (4.5)
ANMS Gastroparesis Cardinal Symptom Index Daily Diary [Mean (Standard Deviation); unit: units on a scale] — American Neurogastroenterology and Motility Society Gastroparesis Cardinal Symptom Index-Daily Diary (ANMS GCSI-DD) has the patient report their gastroparesis symptoms from 0 (none) to 4 (very severe) on a daily basis. The Daily Diary Gastroparesis Cardinal Symptom Index (GCSI-DD) total score is comprised of the average of feeling excessively full after meals and unable to finish a normal size meal, nausea and bloating severity. The baseline score is the average of the 7-days of ANMS GCSI-DD scores during the screening period.
  units on a scale
    Fullness/early satiety subscale | 2.62 (0.94) | 2.68 (0.86) | 2.65 (0.90)
    Early satiety severity | 2.56 (0.78) | 2.59 (0.86) | 2.57 (0.94)
    Excessive fullness severity | 2.40 (0.98) | 2.77 (0.98) | 2.74 (0.94)
PAGI-QOL disease-specific Quality of Life (QOL) Total Score [Mean (Standard Deviation); unit: units on a scale] — Patient Assessment of Upper GastroIntestinal Disorders-Quality of Life (PAGI-QOL), disease-specific QOL questionnaire total score assesses the impact of a patient's disease related to avoiding or having difficulties in the prior 2 weeks due to the patient's gastrointestinal issues rated for 30 items scored from 0 (none) to 5 (all of the time). The total score is the average of 5 domains: Daily Activities, Clothing, Diet and Food Habits, Relationships, and Psychological Well-Being and Distress after reversing item scores so that a low score reflects poor QOL and higher scores reflect high QOL.
  units on a scale | 2.3 (1.1) | 2.4 (1.1) | 2.4 (1.1)
Hospital Anxiety and Depression Scale (HADS) [Mean (Standard Deviation); unit: units on a scale] — The Hospital Anxiety and Depression Scale (HADS) questionnaire is a 14-item scale, that measures 2 subscores: the amount of anxiety, (HADS-A total score) and the level of depression (HADS-D total score), in the prior 2 weeks. Each subscore is 8 items scored from 0 (not at all) to 3 (most of the time) and is computed on a scale of 0 to 21, so that higher scores indicate more severe anxiety or depression.
  units on a scale
    HADS-A total score | 9.3 (4.5) | 9.1 (4.8) | 9.2 (4.6)
    HADS-D total score | 6.7 (5.1) | 6.8 (4.7) | 6.8 (4.9)
SF-36 Quality of Life (QOL) [Mean (Standard Deviation); unit: units on a scale] — The Short-Form 36 v2 is a short-form general health survey that measures each of the following eight health domains: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. Each health domain score contributes to the Physical Component Summary (PCS) and Mental Component Summary (MCS) scores. Each summary score is standardized to range from 0 (very poor QOL) to 100 (excellent QOL).
  units on a scale
    Physical component summary score | 33.7 (8.2) | 33.3 (9.0) | 33.5 (8.6)
    Mental component summary score | 37.9 (15.6) | 41.3 (13.8) | 39.6 (14.7)
Gastric Emptying scintigraphy (GES) [Count of Participants; unit: Participants]
  Not delayed gastric emptying | 20 | 25 | 45
  Delayed gastric emptying | 26 | 22 | 48
  Rapid gastric emptying | 1 | 2 | 3
Intra-gastric meal distribution (IMD) [Count of Participants; unit: Participants] — The Intragastric meal distribution (IMD) is assessed at baseline during the Gastric Emptying Scintigraphy Test. The ratio of gastric counts of the meal in the proximal stomach to the distal stomach is used to compute the Intragastric meal distribution (IMD) which can be used as an indirect measure of Fundic Accommodation. Population: A total of 32 of the 96 patients randomized did not have evaluable data required for the analysis of the intra-gastric meal distribution (16 Buspirone, 16 Placebo patients).
  Participants
    number analyzed (Participants) | 31 | 33 | 64
    Normal (0.644 - 1.00) | 27 | 25 | 52
    Borderline (0.568 - 0.643) | 0 | 3 | 3
    Impaired (<0.568) | 4 | 5 | 9
Water load test, volume consumed [Median (Standard Deviation); unit: mL] | 415.9 (217.0) | 401.7 (198.0) | 408.5 (206.3)
Water load test, consumed low volume (<238 mL) [Count of Participants; unit: Participants] | 9 | 10 | 19

OUTCOME MEASURES:

1. Primary Outcome: 4-Week Change in the Postprandial Fullness and Early Satiety Symptoms Severity
Description: The outcome is assessed using the self-reported early satiety/postprandial fullness subscore (ES/PPF), which is computed as the average of 4 scores for 4-items on the Gastroparesis Cardinal Symptom Index (GCSI) survey: stomach fullness, inability to finish a normal-sized meal, feeling excessively full after meals, and loss of appetite. Each item is scored from 0 (no) to 5 (very severe) symptoms in the past 2-weeks; the subscore ranges from 0 to 5. The change is computed as the subscore at 4-weeks minus the baseline subscore.
Time Frame: baseline and 4-weeks
Population: All participants assigned to the arm with data for the outcome available at 4-weeks.
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 47 | 49
score on a scale | -1.16 (1.25) | -1.03 (1.19)
Statistical Analysis 1: Comparison: Buspirone vs Placebo; Primary outcome analysis uses a difference of differences analysis between Buspirone compared to the Placebo arm in which the adjusted mean difference of differences, Wald 95% Confidence interval and 2-sided P values are determined from a Wald Chi-Square test. Adjusted mean difference of differences (DoD) from baseline were computed using ANCOVA, regressing change from baseline to 4-weeks on treatment group and baseline value of the outcome. Negative change indicates symptom improvement; Test type: Superiority; p = 0.69, ANCOVA — Nominal P value. Power was determined at a level of P=0.05; Multiple imputation using regression and 50 datasets to estimate the outcome for the 18/96 (19%) randomized patients without the f4 visit data; Mean Difference (Net) = -0.11, 95% CI 2-sided [-0.68 to 0.45]
Statistical Analysis 2: Comparison: Buspirone vs Placebo; Sensitivity analysis of change from a baseline in ES/PPF (Early Satiety/Postprandial Fullness subscore) using all completers: 39 participants in Buspirone arm, 39 participants in placebo arm; Test type: Superiority; p = 0.62, ANCOVA — P value is nominal; no adjustments made from multiple comparisons. Bonferroni p-value for the 10 sensitivity outcomes is <0.005; Mean Difference (Net) = -0.13, 95% CI 2-sided [-0.65 to 0.39]
Statistical Analysis 3: Comparison: Buspirone vs Placebo; Sensitivity analyses: change in ES/PPF in treatment adherent patients: 23 participants in Buspirone arm, 29 patients in placebo arm; Test type: Superiority; p = 0.62, ANCOVA — P value is nominal; no adjustments made for multiple comparisons. Bonferroni p-value for the 10 sensitivity outcomes is <0.005; Mean Difference (Net) = -0.25, 95% CI 2-sided [-0.89 to 0.38]

2. Secondary Outcome: 4-Week Change in Stomach Fullness Symptom Severity
Description: The outcome is assessed using self-reported assessment of stomach fullness severity in the prior 2-weeks using the Gastroparesis Cardinal Symptoms Index (GCSI) survey. The item is scored from 0 (no) to 5 (very severe) symptoms; the change is computed as the score at 4-weeks minus the baseline score.
Time Frame: baseline and 4-weeks
Population: All participants assigned to the arm with 4-week visit data
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 47 | 47
score on a scale | -1.16 (1.55) | -1.07 (1.34)
Statistical Analysis 1: Comparison: Buspirone vs Placebo; The mean difference of differences (DoD) between Buspirone and Placebo, 95% confidence interval and P (2-sided) were derived from an ANCOVA, regressing an indicator for treatment group on fullness severity score, adjusting for the baseline value of fullness severity score; Test type: Superiority; p = 0.76, ANCOVA — Nominal P value reported. Bonferroni p-value for the 10 sensitivity outcomes is <0.005; Mean Difference (Net) = -0.09, 95% CI 2-sided [-0.69 to 0.50]

3. Secondary Outcome: 4-Week Change in Excessive Fullness Symptom Severity
Description: The outcome is assessed using self-reported assessment of feeling excessively full after meals severity in the prior 2-weeks using the Gastroparesis Cardinal Symptom Index (GCSI) survey. The item is scored from 0 (no) to 5 (very severe) symptoms; the change is computed as the score at 4-weeks minus the baseline score.
Time Frame: baseline and 4-weeks
Population: All participants assigned to the arm with a 4-week visit and data for excessive fullness severity.
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 39 | 39
score on a scale | -1.14 (1.56) | -0.99 (1.30)
Statistical Analysis 1: Comparison: Buspirone vs Placebo; Adjusted mean difference of differences (DoD) from baseline were computed using ANCOVA, regressing change from baseline to 4-weeks on treatment group and baseline value of the outcome. Wald 95% Confidence Limits (CI) are reported; P (2-sided) determined from a Wald Chi-Square test; Test type: Superiority; p = 0.64, ANCOVA — Nominal P values; Bonferroni p value for the 10 sensitivity outcomes is <0.005; Mean Difference (Net) = -0.15, 95% CI 2-sided [-0.76 to 0.47]

4. Secondary Outcome: 4-Week Change in Inability to Finish a Normal-sized Meal Symptom Severity
Description: The outcome is assessed using self-reported assessment of inability to finish a normal-sized meal severity in the prior 2-weeks using the Gastroparesis Cardinal Symptom Index (GCSI) survey. The item is scored from 0 (no) to 5 (very severe) symptoms; the change is computed as the score at 4-weeks minus the baseline score. A negative change indicates symptom improvement.
Time Frame: baseline and 4-weeks
Population: All participants assigned to the arm with a 4-week visit.
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 39 | 39
score on a scale | -1.27 (1.55) | -1.12 (1.63)
Statistical Analysis 1: Comparison: Buspirone vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.66, ANCOVA — P values are nominal; Bonferroni p-value for the 10 sensitivity outcomes is <0.005; Mean Difference (Net) = -0.14, 95% CI 2-sided [-0.79 to 0.50]

5. Secondary Outcome: 4-Week Change in Loss of Appetite Symptom Severity
Description: The outcome is assessed using self-reported assessment of loss of appetite severity in the prior 2-weeks using the Gastroparesis Cardinal Symptom Index (GCSI) survey. The item is scored from 0 (no) to 5 (very severe) symptoms; the change is computed as the score at 4-weeks minus the baseline score. A negative change indicates symptom improvement.
Time Frame: baseline and 4-weeks
Population: All participants assigned to the arm with a 4-week visit and values for loss of appetite severity.
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 39 | 39
score on a scale | -1.09 (1.64) | -0.96 (1.62)
Statistical Analysis 1: Comparison: Buspirone vs Placebo; Adjusted mean difference of differences (DoD) from baseline were computed using ANCOVA, regressing change from baseline to 4-weeks on treatment group and baseline value of the outcome. Wald 95% Confidence Limits (CI) are reported; P (s-sided) determined from a Wald Chi-Square test; Test type: Superiority; p = 0.70, ANCOVA — Nominal P values; Bonferroni p-value for the 10 sensitivity outcomes is <0.005; Mean Difference (Net) = -0.12, 95% CI 2-sided [-0.75 to 0.50]

6. Secondary Outcome: 4-Week Change in Total Overall GCSI Symptom Severity
Description: The outcome is assessed using the self-reported Gastroparesis Cardinal Symptom Index (GCSI) total score, which is computed as the average of the 3 subscores on the GCSI survey: 3-item early satiety/postprandial fullness subscore, the nausea/vomiting subscore (average of 3-items: nausea, retching, vomiting), and bloating subscore (average of 2-items: bloating, stomach visibly larger). Each item is scored from 0 (no) to 5 (very severe) symptoms in the past 2-weeks; the total score ranges from 0 to 5. The change is computed as the total score at 4-weeks minus the baseline total score. A negative change indicates improved symptoms.
Time Frame: baseline and 4-weeks
Population: All patients with 4-week visit data for GCSI.
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 39 | 39
score on a scale | -1.06 (1.16) | -0.86 (1.00)
Statistical Analysis 1: Comparison: Buspirone vs Placebo; Adjusted mean difference of differences (DoD) of change in outcome from baseline and 95% Confidence Intervals were computed using ANCOVA, regressing change from baseline to 4-weeks on treatment group and baseline value of the outcome. P (2-sided) were determined from a Wald Chi-Square test; Test type: Superiority; p = 0.40, ANCOVA — P value is nominal; no adjustments made for multiple comparisons. Bonferrini p-value is <0.002; Mean Difference (Net) = -0.20, 95% CI 2-sided [-0.66 to 0.27]
Statistical Analysis 2: Comparison: Buspirone vs Placebo; GCSI symptomatic improvement of 1+ points in total GCSI symptom score defined as change in GCSI total score at week 4 from baseline being a decrease of 1 or more points. This is a binary variable where 1=1+ reduction in change in GCSI total score, 0=change in GCSI total score from baseline at 4-weeks is < 1.0; Test type: Superiority; p = 0.56, Regression, Logistic — Nominal P value without adjustment for multiple comparisons. Bonferroni threshold for level of significance is <0.002; Odds ratio, 95% C.I. and P (two-sided) from a logistic regression of the binary outcome on treatment group for symptomatic improvement in GCSI; Odds Ratio (OR) = 1.31, 95% CI 2-sided [0.53 to 3.21]

7. Secondary Outcome: 4-Week Change in Nausea, Vomiting and Retching Symptoms Severity
Description: The outcome is assessed using the self-reported nausea/vomiting subscore, which is computed as the average of 3 scores for 3-items on the Gastrointestinal Cardinal Symptom Index (GCSI) survey: nausea, retching, vomiting. Each item is scored from 0 (no) to 5 (very severe) symptoms in the past 2-weeks. The change is computed as the subscore at 4-weeks minus the baseline subscore. Negative change indicates improvement in symptoms.
Time Frame: baseline and 4-weeks
Population: All participants assigned to the arm with a 4-week visit and data for the nausea/vomiting subscore.
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 39 | 39
score on a scale | -0.65 (1.40) | -0.60 (1.26)
Statistical Analysis 1: Comparison: Buspirone vs Placebo; Adjusted mean difference of differences (DoD) from baseline were computed using ANCOVA, regressing change from baseline to 4-weeks on treatment group and baseline value of the outcome. Wald 95% Confidence Limits (CI) are reported; P (2-sided) determined from a Wald Chi-Squares test; Test type: Superiority; p = 0.86, ANCOVA — P value is nominal: no adjustments made for multiple comparisons. Bonferroni p-value threshold for the level of significance is <0.002; Mean Difference (Net) = -0.05, 95% CI 2-sided [-0.58 to 0.48]

8. Secondary Outcome: 4-Week Change in Nausea Symptom Severity
Description: The outcome is assessed using self-reported assessment of nausea severity item from the Patient Assessment of Upper Gastrointestinal Disorders Symptom Severity Index (PAGI-SYM) in the prior 2-weeks using the Gastroparesis Cardinal Symptom Index (GCSI) survey. The item is scored from 0 (no) to 5 (very severe) symptoms; the change is computed as the score at 4-weeks minus the baseline score.
Time Frame: baseline and 4-weeks
Population: All participants assigned to the arm with a 4-week visit and data for the nausea severity.
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 39 | 39
score on a scale | -0.75 (1.40) | -0.70 (1.51)
Statistical Analysis 1: Comparison: Buspirone vs Placebo; Adjusted mean difference of differences (DoD) from baseline were computed using ANCOVA, regressing change from baseline to 4-weeks on treatment group and baseline value of outcome. Wald 95% Confidence Limits (CI) are reported; P (2-sided) determined from a Wald-Chi Square test; Test type: Superiority; p = 0.85, ANCOVA — P value is nominal; no adjustments made for multiple comparisons. Bonferroni p-value is <0.002; Mean Difference (Net) = -0.06, 95% CI 2-sided [-0.64 to 0.53]

9. Secondary Outcome: 4-Week Change in Vomiting Symptom Severity
Description: The outcome is assessed using self-reported assessment of vomiting severity in the prior 2-weeks using the Gastroparesis Cardinal Symptom Index (GCSI) survey. The item is scored from 0 (no) to 5 (very severe) symptoms; the change is computed as the score at 4-weeks minus the baseline score. A negative change indicates improvement in vomiting severity.
Time Frame: baseline and 4-weeks
Population: All participants assigned to the arm with a 4-week visit and data for vomiting severity.
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 39 | 39
score on a scale | -0.71 (1.81) | -0.57 (1.47)
Statistical Analysis 1: Comparison: Buspirone vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.65, ANCOVA — P value is nominal; no adjustments made for multiple comparisons. Bonferroni p-value is <0.002; Mean Difference (Net) = -0.14, 95% CI 2-sided [-0.76 to 0.47]

10. Secondary Outcome: 4-Week Change in Bloating and Stomach Distention Symptoms Severity
Description: The outcome is assessed using the self-reported bloating subscore, which is computed as the average of 2 scores for 2-items on the Gastroparesis Cardinal Symptom Index (GCSI) survey: bloating, stomach visibly larger. Each item is scored from 0 (no) to 5 (very severe) symptoms in the past 2-weeks; the subscore ranges from 0 to 5. The change is computed as the subscore at 4-weeks minus the baseline subscore. A negative value for change indicates improvement in symptoms.
Time Frame: baseline and 4-weeks
Population: All participants assigned to the arm with a 4-week visit data for the bloating subscore.
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 39 | 39
score on a scale | -1.36 (1.42) | -0.95 (1.27)
Statistical Analysis 1: Comparison: Buspirone vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.16, ANCOVA — P value is nominal: no adjustments made for multiple comparisons. Bonferroni p-value threshold level of significance is <0.002; Mean Difference (Net) = -0.41, 95% CI 2-sided [-0.99 to 0.16]

11. Secondary Outcome: 4-Week Change in Bloating Symptom Severity
Description: The outcome is assessed using self-reported assessment of bloating severity in the prior 2-weeks using the Gastroparesis Cardinal Symptom Index (GCSI) survey. The item is scored from 0 (no) to 5 (very severe) symptoms; the change is computed as the score at 4-weeks minus the baseline score. A negative change indicates symptom improvement.
Time Frame: baseline and 4-weeks
Population: All participants assigned to the treatment arm with a 4-week visit and data for bloating severity.
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 39 | 39
score on a scale | -1.34 (1.46) | -0.69 (1.18)
Statistical Analysis 1: Comparison: Buspirone vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.03, ANCOVA — P values are nominal; no adjustments made for multiple comparisons; Mean Difference (Net) = -0.65, 95% CI 2-sided [-1.23 to -0.08]

12. Secondary Outcome: 4-Week Change in Upper Abdominal Pain and Discomfort Symptoms Severity
Description: The outcome is assessed using the self-reported upper abdominal pain subscore, which is computed as the average of 2 scores for 2-items on the Patient Assessment of Upper Gastrointestinal Disorders-Symptom Severity Index (PAGI-SYM) survey: upper abdominal pain, upper abdominal discomfort. Each item is scored from 0 (no) to 5 (very severe) symptoms in the past 2-weeks; the subscore ranges from 0 to 5. The change is computed as the subscore at 4-weeks minus the baseline subscore.
Time Frame: baseline and 4-weeks
Population: All participants assigned to the arm with a 4-week visit and values for the upper abdominal pain subscore.
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 39 | 39
score on a scale | -0.78 (1.55) | -0.95 (1.63)
Statistical Analysis 1: Comparison: Buspirone vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.59, ANCOVA — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = 0.17, 95% CI 2-sided [-0.44 to 0.77]

13. Secondary Outcome: 4-Week Change in Upper Abdominal Pain Symptom Severity
Description: The outcome is assessed using self-reported assessment of upper abdominal pain severity in the prior 2-weeks using the Patient Assessment of Upper Gastrointestinal Disorders Symptom Severity Index (PAGI-SYM) survey. The item is scored from 0 (no) to 5 (very severe) symptoms; the change is computed as the score at 4-weeks minus the baseline score. A negative change indicates symptom improvement.
Time Frame: baseline and 4-weeks
Population: All participants assigned to the arm with a 4-week visit and upper abdominal pain severity data.
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 39 | 39
score on a scale | -0.69 (1.73) | -0.93 (1.63)
Statistical Analysis 1: Comparison: Buspirone vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.46, ANCOVA — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = 0.24, 95% CI 2-sided [-0.39 to 0.88]

14. Secondary Outcome: 4-Week Change in Gastroesophageal (GERD) Symptoms Severity
Description: The outcome is assessed using the self-reported GERD subscore, which is computed as the average of 7 scores for 7-items on the Patient Assessment of Gastrointestinal Disorders Symptom Severity Index (PAGI-SYM) survey: heartburn during the day, heartburn when lying down, feeling of discomfort inside chest during the day, feeling of discomfort inside chest during sleep, regurgitation or reflux during the day, regurgitation when lying down, bitter, acid or sour taste in mouth. Each item is scored from 0 (no) to 5 (very severe) symptoms in the past 2-weeks; the subscore ranges from 0 to 5. The change is computed as the subscore at 4-weeks minus the baseline subscore.
Time Frame: baseline and 4-weeks
Population: All participants assigned to the arm with 4-week visit data for the GERD subscore.
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 38 | 39
score on a scale | -0.36 (1.44) | -0.45 (1.01)
Statistical Analysis 1: Comparison: Buspirone vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.73, ANCOVA — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = 0.09, 95% CI 2-sided [-0.42 to 0.59]

15. Secondary Outcome: 4-Week Change in Gastrointestinal Symptoms Rating Scale (GSRS) Global Score
Description: The outcome is assessed using the self-reported GSRS total score which is computed as the mean of the 15 item scores on the Gastrointestinal Symptom Rating Scale (GSRS) survey. Each item is scored from 1 (no discomfort) to 7 (very severe discomfort) of the symptom in the past week. The change is computed as the score at 4-weeks minus the baseline score. A negative change indicates symptom improvement.
Time Frame: baseline and 4-weeks
Population: All participants assigned to the arm with a 4-week visit and data for the GSRS total score.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 39 | 38
units on a scale | -0.63 (1.09) | -0.49 (0.90)
Statistical Analysis 1: Comparison: Buspirone vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.50, ANCOVA — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = -0.14, 95% CI 2-sided [-0.55 to 0.27]

16. Secondary Outcome: 4-Week Change in Participant's Rating of Symptom Relief
Description: The outcome is assessed using the participant-rated Clinical Patient Grading Assessment Scale (CPGAS) score which is scored from -3 (very considerably worse) to 3 (completely better) in the past week compared to the way the participant usually feels. The change is computed as the score at 4-weeks minus the baseline score. A positive change indicates patient feeling better.
Time Frame: baseline and 4-weeks
Population: All participants assigned to the arm with a 4-week visit and data for CPGAS score.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 39 | 39
units on a scale | 0.69 (1.03) | 0.37 (1.10)
Statistical Analysis 1: Comparison: Buspirone vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.18, ANOVA — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = 0.32, 95% CI 2-sided [-0.15 to 0.79]

17. Secondary Outcome: 4-Week Change in Severity of Somatic Symptoms
Description: The outcome is assessed using the self-reported Patient Health Questionnaire 15 Somatic Symptom Severity Scale (PHQ-15) total somatization score (ranges from 0 -30, with 30 being most bothered by symptoms in prior 4-weeks), calculated as the sum of 15-items, each scored from 0 (not bothered at all) to 2 (bothered a lot) by somatic symptoms in the prior 4-weeks. The change is computed as the score at 4-weeks minus the baseline score. A negative change indicates being less bothered by the symptoms.
Time Frame: baseline and 4-weeks
Population: Participants in each arm with the total somatization score at 4-weeks.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 39 | 39
units on a scale | -0.99 (3.88) | -2.00 (3.93)
Statistical Analysis 1: Comparison: Buspirone vs Placebo; Adjusted mean difference from differences (DoD) from the baseline were computed using ANCOVA, regressing change from baseline to 4-weeks on treatment group and baseline value of the outcome. Wald 95% Confidence Intervals are reported; P value (2-sided) determined from a Wald Chi-Square test; Test type: Superiority; p = 0.19, ANCOVA — P value is nominal: no adjustments made from multiple comparisons. Bonferroni p-value threshold for the level of significance is <0.002; Mean Difference (Net) = 1.01, 95% CI 2-sided [-0.49 to 2.51]

18. Secondary Outcome: 4-Week Change in Depression
Description: The outcome is assessed using the self-reported Hospital Anxiety and Depression Scale (HADS) depression subscore, calculated as the sum of 7 items, each scored from 0 (not at all) to 3 (most of the time). The change is computed as the subscore at 4-weeks minus the baseline subscore. A negative change indicates reduced depression.
Time Frame: baseline and 4-weeks
Population: Participants in each arm with HADS data at 4-weeks. 1 Placebo patient did not have HADS data at 4-weeks.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 39 | 38
units on a scale | 0.42 (4.06) | -1.43 (3.91)
Statistical Analysis 1: Comparison: Buspirone vs Placebo; Adjusted mean difference of differences (DoD) from baseline were computed using ANCOVA, regressing change from baseline to 4-weeks on treatment group and baseline value of the HADS depression score; Test type: Superiority; p = 0.02, ANCOVA — P value is nominal: no adjustments made for multiple comparisons. Bonferroni P-value threshold for the level of significance is <=0.002; Mean Difference (Net) = 1.86, 95% CI 2-sided [0.33 to 3.38]

19. Secondary Outcome: 4-Week Change in Anxiety
Description: The outcome is assessed using the self-reported Hospital Anxiety and Depression Scale (HADS) anxiety subscore, calculated as the sum of 7-items, each scored from 0 (not at all) to 3 (most of the time). The change is computed as the subscore at 4-weeks minus the baseline subscore. A negative change indicates reduced anxiety at 4-weeks.
Time Frame: baseline and 4-weeks
Population: Participants in each arm with HADS anxiety data at 4-weeks. 1 Placebo patient did not report a HADS anxiety subscale score at 4 -weeks.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 39 | 38
units on a scale | -1.27 (4.82) | -2.03 (3.94)
Statistical Analysis 1: Comparison: Buspirone vs Placebo; Adjusted mean difference of differences (DoD) from baseline were computed using ANCOVA, regressing change from baseline to 4-weeks on treatment group and baseline value of the HADS anxiety total score. 95% Wald Confidence Intervals are reported; P (2-sided) determined from a Wald Chi-Square test; Test type: Superiority; p = 0.40, ANCOVA — P values are nominal; no adjustments for multiple comparisons; Mean Difference (Net) = 0.76, 95% CI 2-sided [-1.02 to 2.54]

20. Secondary Outcome: 4-Week Change Overall Quality of Health Due to Gastroparesis Issues
Description: The outcome is assessed using the self-reported Patient Assessment of Upper Gastrointestinal Disorders-Quality of Life (PAGI-QOL) total score which comprises 30 items scored from 0 (none of the time) to 5 (all of the time) the participant's QOL has been affected by their gastrointestinal issues in the prior two weeks. The total score is the mean of the 5 subscale scores and ranges from 0 (lowest QOL) to 5 (highest QOL) in past 2-weeks. The change is computed as the score at 4-weeks minus the baseline score. A positive change indicates improved QOL.
Time Frame: baseline and 4-weeks
Population: Participants with available PAGI-QOL data at 4-weeks. 1 Placebo patient did not have values for PAGI-QOL total score.
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 39 | 38
score on a scale | 0.43 (0.81) | 0.64 (0.95)
Statistical Analysis 1: Comparison: Buspirone vs Placebo; Adjusted mean difference of differences (DoD) from baseline were computed using ANCOVA, regressing change from baseline to 4-weeks on treatment group and baseline value of PAGI-QOL total score; Test type: Superiority; p = 0.25, ANCOVA — P value is nominal with no adjustment for multiple comparisons. The Bonferroni level of significance threshold is <=0.002; Mean Difference (Net) = -0.21, 95% CI 2-sided [-0.57 to 0.15]

21. Secondary Outcome: 4-Week Change in Overall Mental Quality of Life (QOL)
Description: The outcome is assessed using the self-reported 36-item Short Form Health Survey (SF-36v2) mental health QOL component score. The score ranges from 0 (poorest) to 100 (highest) QOL. The change is computed as the score at 4-weeks minus the baseline score. A positive change indicates improved mental QOL.
Time Frame: baseline and 4-weeks
Population: All participants in the treatment arm with baseline and mental QOL data at 4-weeks.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 39 | 39
units on a scale | 1.19 (10.54) | 3.17 (11.83)
Statistical Analysis 1: Comparison: Buspirone vs Placebo; Adjusted mean difference of differences (DoD) of change in outcome from baseline and 95% Confidence Intervals were computed using ANCOVA, regressing change from baseline to 4-weeks on treatment group and baseline value of outcome. P (2-sided) were determined from a Wald-Chi-Square test; Test type: Superiority; p = 0.36, ANCOVA; Mean Difference (Net) = -1.98, 95% CI 2-sided [-6.20 to 2.24]

22. Secondary Outcome: 4-Week Change in Overall Physical Quality of Life (QOL)
Description: The outcome is assessed using the self-reported 36-item Short Form Health Survey (SF-36v2) physical health QOL component score. The score ranges from 0 (poorest) to 100 (highest) QOL. The change is computed as the score at 4-weeks minus the baseline score. A positive change indicates improved Physical QOL.
Time Frame: baseline and 4-weeks
Population: All participants assigned to the arm with a 4-week visit and data for the Physical QOL summary score.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 39 | 39
units on a scale | 1.10 (7.18) | 3.17 (5.95)
Statistical Analysis 1: Comparison: Buspirone vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.15, ANCOVA — P value is nominal; no adjustments made for multiple comparisons Bonferroni p-value is <0.002; Mean Difference (Net) = -2.07, 95% CI 2-sided [-4.91 to 0.76]

23. Secondary Outcome: 4-Week Change in Gastric Retention
Description: The outcome is assessed using the percent of gastric retention at 4-hours from the Gastric Emptying Scintigraphy (GES) test. The change is computed as the percent retention at 4-weeks minus the baseline percent retention. % retention is the amount of food remaining in the stomach at 4-hours of the GES test and ranges from 0% (no food) to 100% (all of the food).
Time Frame: baseline and 4-weeks
Population: All participants assigned to the arm that had 4 week visit data for the GES test at 4-hours.
Measure: Least Squares Mean (Standard Deviation); unit: units on a percentage scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 26 | 33
units on a percentage scale | 4.24 (21.19) | 2.87 (21.8)
Statistical Analysis 1: Comparison: Buspirone vs Placebo; Adjusted mean difference of differences (DoD) from baseline were computed using ANCOVA regressing change from baseline to 4-weeks on treatment group and baseline value of the outcome. Wald 95% Confidence Intervals are reported. P (2-sided) determined from a Wald Chi-Square test; Test type: Superiority; p = 0.76, ANCOVA — P value is nominal: no adjustments made for multiple comparisons. Bonferrini p-value is <0.002; Mean Difference (Net) = 1.37, 95% CI 2-sided [-7.51 to 10.25]

24. Secondary Outcome: Change at 4-weeks in the Intragastric Meal Distribution (IMD)
Description: The Intragastric meal distribution (IMD) is assessed at baseline and 4-weeks during the Gastric Emptying Scintigraphy Test. The ratio of gastric counts of the meal in the proximal stomach to the distal stomach is used to compute the Intragastric meal distribution (IMD) which can be used as an indirect measure of Fundic Accommodation.
Time Frame: baseline and 4-weeks
Population: Patients in each treatment arm with measurements for IMD at 4-weeks.
Measure: Least Squares Mean (Standard Deviation); unit: ratio
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 17 | 24
ratio | -0.04 (0.13) | 0.02 (0.13)
Statistical Analysis 1: Comparison: Buspirone vs Placebo; Adjusted mean difference of differences (DoD) were computed using ANCOVA, regressing change in IMD from baseline to 4-weeks on treatment group and the baseline value of IMD. Wald 95% Confidence Intervals are reported; P (2-sided) determined from a Wald Chi-Square test; Test type: Superiority; p = 0.10, ANCOVA — Nominal P values; no adjustment for multiple comparisons; Mean Difference (Net) = -0.05, 95% CI 2-sided [-0.12 to 0.01]

25. Secondary Outcome: Change From Baseline at 4-weeks in the Water Load Satiety Test (WLST)
Description: The Water Load Satiety Test (WLST) is the amount of water a patient can consume until full in 5 minutes. The volume of water is recorded. The change is computed as the volume of water ingested at baseline subtracted from the amount of water ingested at 4-weeks. A positive change indicates that the patient can ingest more water at 4-weeks than at baseline.
Time Frame: baseline and 4-weeks
Population: Participants in each treatment arm with a volume of water measured at both baseline and 4-weeks.
Measure: Least Squares Mean (Standard Error); unit: ml
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 26 | 26
ml | -43.3 (219.1) | -21.8 (145.6)
Statistical Analysis 1: Comparison: Buspirone vs Placebo; Adjusted mean difference of differences (DoD) from baseline were computed using ANCOVA, regressing change from baseline to 4-weeks on treatment group and baseline value of teh outcome. Wald 95% Confidence Limits are reported; P (2-sided) determined from a Wald Chi-Square test; Test type: Superiority; p = 0.29, ANCOVA — Nominal P values; no adjustments for multiple comparisons; Mean Difference (Net) = -21.51, 95% CI 2-sided [-99.4 to 56.4]

26. Other Pre Specified Outcome: 4-Week Change in Weight
Description: This safety outcome is computed by subtracting the weight (kg) at baseline from the weight (kg) at 4-weeks
Time Frame: baseline and 4-weeks
Population: All participants assigned to the arm with a 4-week visit and a measurement for weight.
Measure: Least Squares Mean (Standard Deviation); unit: kilogram
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 26 | 29
kilogram | -0.34 (1.36) | -0.43 (1.99)
Statistical Analysis 1: Comparison: Buspirone vs Placebo; Adjusted mean difference of differences (DoD) from baseline were computed using ANCOVA, regressing change from baseline to week 4 on treatment group and baseline value of the outcome. Wald 95% Confidence Limits (CI) are reported: P (2-sided) determined from Wald Chi-Square test; Test type: Superiority; p = 0.84, ANCOVA — P value is nominal; no adjustments made for multiple comparisons. Bonferroni p-value <0.002; Mean Difference (Net) = 0.09, 95% CI 2-sided [-0.78 to 0.95]

27. Other Pre Specified Outcome: 4-Week Cardiac Rhythm
Description: This safety outcome is computed from the results of an electrocardiogram (ECG) QTc interval at 4-weeks measured in milliseconds (msec).
Time Frame: baseline and 4-weeks
Population: All participants assigned to the arm with 4-week visit data for the Electrocardiogram QTc interval.
Measure: Least Squares Mean (Standard Deviation); unit: milliseconds (msec)
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 26 | 29
milliseconds (msec) | -2.80 (19.18) | 3.63 (23.42)
Statistical Analysis 1: Comparison: Buspirone vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.27, ANCOVA — P value is nominal; Mean Difference (Net) = -6.43, 95% CI 2-sided [-17.90 to 5.03]

28. Other Pre Specified Outcome: 4-Week Change in Aspartate Aminotransferase (ALT)
Description: This safety outcome is computed by subtracting the baseline level of Alanine Aminotransferase (ALT) (U/L) from the 4-week level.
Time Frame: baseline and 4-weeks
Population: All participants assigned to the arm with a 4-week visit and a measurement for ALT.
Measure: Least Squares Mean (Standard Deviation); unit: U/L
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 28 | 33
U/L | 0.32 (15.93) | 1.34 (9.57)
Statistical Analysis 1: Comparison: Buspirone vs Placebo; Adjusted mean difference of differences (DoD) from baseline were computed using ANCOVA, regressing change from baseline to 4-weeks on treatment group and baseline value of the outcome. Wald 95% Confidence Intervals are reported; P (2-sided) determined from a Wald Chi-Square test; Test type: Superiority; p = 0.74, ANCOVA — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = -1.02, 95% CI 2-sided [-6.93 to 4.89]

29. Other Pre Specified Outcome: 4-Week Change in Creatinine
Description: This safety outcome is computed by subtracting the baseline level of creatinine (mg/dL) from the 4-week level.
Time Frame: baseline and 4-weeks
Population: All participants assigned to the arm with a 4-week visit and a measurement for Creatinine.
Measure: Least Squares Mean (Standard Deviation); unit: mg/dL
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 27 | 33
mg/dL | 0.02 (0.07) | -0.01 (0.11)
Statistical Analysis 1: Comparison: Buspirone vs Placebo; Adjusted mean difference of differences (DoD) from baseline were computed using ANCOVA, regressing change from baseline to 4-weeks on treatment group and baseline value of the outcome. 95% Wald Confidence Intervals are reported; P (2-sided) determined from a Wald Chi-Square test; Test type: Superiority; p = 0.18, ANCOVA; P value is nominal: no adjustments made for multiple comparisons. Bonferroni p-value threshold level of significance <0.002; Mean Difference (Net) = 0.03, 95% CI 2-sided [-0.01 to 0.08]

30. Other Pre Specified Outcome: 4-Week Change in Fasting Glucose
Description: This safety outcome is computed by subtracting the baseline level of glucose (mg/dL) from the 4-week level.
Time Frame: baseline and 4-weeks
Population: All participants assigned to the arm with a 4-week visit with a measurement for glucose.
Measure: Least Squares Mean (Standard Deviation); unit: mg/dL
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 27 | 33
mg/dL | 10.30 (38.10) | 10.69 (42.21)
Statistical Analysis 1: Comparison: Buspirone vs Placebo; [analysis description as in outcome 29, analysis 1]; Test type: Superiority; p = 0.97, ANCOVA — [p-value comment as in outcome 10, analysis 1]; Mean Difference (Net) = -0.39, 95% CI 2-sided [-20.42 to 19.64]

31. Other Pre Specified Outcome: Assessment of Adverse Events Over 4-Weeks
Description: This safety outcome is the frequency over the 4-weeks of the study of all reported adverse events using the v5.0 CTCAE classification system.
Time Frame: over 4-weeks
Measure: Number; unit: events
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 47 | 49
events | 12 | 8
Statistical Analysis 1: Comparison: Buspirone vs Placebo; Event rates are computed by treatment arm by dividing the total adverse events over 4-weeks by the number of patient-months of follow-up to 4-weeks. Event rates are compared by treatment arm using an exact poisson regression for event rates; Test type: Superiority; p = 0.64, Exact poisson regression — P values are nominal and not adjusted for multiple comparisons; Incident rate ratio = 1.27, 95% CI 2-sided [0.57 to 2.82]

32. Other Pre Specified Outcome: Assessment of the Severity of Adverse Events Over 4-Weeks
Description: This safety outcome is the frequency over the 4-weeks of the study of all reported adverse events' severity grade as classified by the NCI's Common Terminology Criteria for Adverse Events (CTCAE v5.0). For the patient with 2 AE's, the AE with the maximum severity is reported.
Time Frame: over 4-weeks
Population: All participants randomized in the trial with events occurring over the 4 weeks of follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 47 | 49
Participants
  No Adverse events | 35 | 41
  1-mild severity | 5 | 2
  2-moderate severity | 6 | 6
  3-severe | 1 | 0
  4-life threatening | 0 | 0
  5-death | 0 | 0
Statistical Analysis 1: Comparison: Buspirone vs Placebo; A Fisher's Exact test was used for comparisons of events by treatment by severity grade. One patient in the Buspirone arm had 2 AEs during the trial; for analysis by severity grade the maximum severity grade was used; Test type: Superiority; p = 0.54, Fisher Exact — P values are nominal; Incident rate ratio = 0.95, 95% CI 2-sided [0.35 to 2.62]; An exact poisson regression stratified by severity level was used to compute the incident rate ratio and 95% Confidence Intervals for adverse events by severity level

33. Other Pre Specified Outcome: Serious Adverse Events
Description: Serious Adverse Event (SAE) defined by the FDA as an event meeting one or more of the following criteria; inpatient hospitalization or prolonged existing hospitalization; persistent or significant incapacity or substantial disruption of ability to conduct normal life functions; jeopardized patient and required medical or surgical intervention to prevent a serious event; or congenital anomaly or birth defect.
Time Frame: over 4 weeks of treatment
Population: All patients randomized into each treatment arm
Measure: Number; unit: Serious adverse events
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 47 | 49
Serious adverse events | 1 | 1
Statistical Analysis 1: Comparison: Buspirone vs Placebo; Test type: Superiority; p = 1.00, Fisher Exact — P value is nominal

34. Other Pre Specified Outcome: Total Number of Hospitalizations Over 4-weeks of Treatment
Description: Hospitalization events by treatment arm were reported on the Adverse Event Case-Report form at each visit and also at time of occurrence and tabulated at end of treatment visit for comparison between placebo and buspirone arms.
Time Frame: over the 4-weeks of the trial
Population: all participants by treatment arm randomized into the trial
Measure: Number; unit: hospitalizations
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 47 | 49
hospitalizations | 1 | 0
Statistical Analysis 1: Comparison: Buspirone vs Placebo; Event rates were computed by dividing the number of hospitalizations over 4-weeks by the number of person-years. An exact poisson regression was used to compare events by treatment group; Test type: Superiority; p = 1.00, Exact poisson regression — P-values are nominal; Incident rate ratio = 1.03, 95% CI 2-sided [0 to 40.36]

35. Other Pre Specified Outcome: Adverse Events by Body Classification System by Treatment Group During the Trial
Description: Adverse events were reported on the Adverse Event Report form by the principal investigator at each clinic site using the CTCAE v5 classification system.
Time Frame: over 4-weeks of treatment
Population: All patients randomized into each treatment group.
Measure: Number; unit: events by body classification
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 47 | 49
events by body classification
  Gastrointestinal | 3 | 3
  Immune system | 1 | 0
  Infections & infestations | 3 | 1
  Investigations | 0 | 2
  Metabolic & nutrition | 1 | 0
  Nervous system | 3 | 0
  Renal & urinary | 1 | 1
  Surgical & medical | 0 | 1
  Musculoskeletal & connective tissue disorders | 0 | 1
  Total | 12 | 9
Statistical Analysis 1: Comparison: Buspirone vs Placebo; Test type: Superiority; p = 0.52, Binomial probability test — Nominal P value; 2-sided test with probability of success=0

ADVERSE EVENTS:
Time Frame: Adverse events were counted after randomization through end of treatment at 4-weeks.
Description: Adverse events coded for severity grade using the NCI's Common Terminology Criteria for Adverse Events (v5.0 CTCAE).
Arm/Group | Buspirone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/49
Serious Adverse Events (participants affected / at risk) | 1/47 | 1/49
Other Adverse Events (participants affected / at risk) | 11/47 | 7/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Buspirone (N=47) | Placebo (N=49)
neurostimulator implantation (Surgical and medical procedures) | 0 (0) | 1 (1) — Neurostimulator implantation (elective surgery) occurred at week 2, event judged not related to treatment
severe allergic reaction (Immune system disorders) | 1 (1) | 0 (0) — Patient on Buspirone had severe allergic reaction to mannitol with her other drugs at week 2 resulting in significant incapacity with normal life function; judged definitely not related to treatment, severity grade=3
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Buspirone (N=47) | Placebo (N=49)
Nausea, vomiting, retching (Gastrointestinal disorders) | 3 (3) | 2 (3)
upper respiratory & sinus infection (Infections and infestations) | 3 (3) | 1 (1)
QTC interval was high (Investigations) | 0 (0) | 2 (2)
Worsening of a comorbid illness (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Episodes of dizziness and somnolence (Nervous system disorders) | 3 (3) | 0 (0)
urinary tract infection & renal calculi (Renal and urinary disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Pain in extremity from injured ligament

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-13): https://cdn.clinicaltrials.gov/large-docs/42/NCT03587142/Prot_SAP_000.pdf
  • Informed Consent Form (2021-09-15): https://cdn.clinicaltrials.gov/large-docs/42/NCT03587142/ICF_001.pdf